CLINICAL TRIAL: NCT02654795
Title: AssesSment of the Left Atrial Appendage morphoLogy in Patients aAfter ischeMic Stroke
Brief Title: Assessment of Left Atrial Appendage Morphology in Patients After Ischemic Stroke
Acronym: ASSAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Jakub Baran MD PhD, Principal Investigator, Centre of Postgraduate Medical Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 501-1-10-14-13
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients without stroke (Placebo Comparator): This group will consists of patients scheduled for atrial fibrillation ablation without history of stroke.
  Interventions: Radiation: computed tomography
- Patients with history of stroke (Experimental): This group will consists of patients after ischemic stroke and history of atrial fibrillation.
  Interventions: Radiation: computed tomography

INTERVENTIONS:
Radiation: computed tomography — CT angiography will be performed with a dual-source CT scanner using prospective ECG gating, with detector collimation of 128x0.6 mm, a gantry rotation time of 280 ms, tube voltage of 100-120 kV, tube current of 280-380 mAs depending on the patient's body mass.

SUMMARY:
Stroke remains the most dangerous and frightening complication of atrial fibrillation (AF). Numerous factors predisposing to peripheral embolism in patients with AF have been well defined, documented and included in the CHA2DS2VASC score. Although proper anticoagulation minimizes the risk attributable to "known" risk factors, stroke may still occur. Thus, "unknown" risk factors may play an important role in stroke risk stratification in patients with AF. The investigators assume that one of the important "unknown" risk factor is left atrial appendage (LAA) morphology. The ASSAM study is planned to include 100 patients after ischemic stroke or transient ischemic attack (TIA) and known status of anticoagulation at the time of stroke. The control group will consist of 100 patients scheduled for AF ablation without a history of stroke or TIA.

ELIGIBILITY:
Inclusion Criteria:

* history of ischemic stroke or transient ischemic attack
* history of AF/AL
* known status of anticoagulation at the time of stroke (treatment dose, INR level)

Exclusion Criteria:

* hemorrhagic stroke
* serious renal impairment with GFR <30 ml/min
* hyperthyroidism
* allergy to the contrast agent
* mental inability to sign the informed consent
* receptive aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The LAA morphology in patients with an elevated risk of peripheral thromboembolism defined as CHA2DS2-VAScore >2 | Through study completion, an average of 1 year
  The investigators will examine association of specific type of LAA morphology with ischemic stroke taking in to account anticoagulation in the time of stroke/TIA.
  The morphology of LAA will be divided into 4 types:
  * the chicken wing - LAA with only one lobe, its length exceeds 40 mm and its bend angle is less than 100 degrees
  * the windsock - LAA with one dominant lobe (length > 40 mm) and several secondary, or even tertiary ones, its length exceeds 40 mm and its bend angle exceeds 100 degrees
  * the cauliflower - LAA with a variable number of lobes with lack of a dominant lobe, its total length is less than 40 mm
  * the cactus - LAA with a dominant central lobe with several secondary ones, its total length less than 40 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Grenadierow 51/59, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No